CLINICAL TRIAL: NCT04969939
Title: Investigation of Efficacy and Safety of NNC0165-1875 as add-on to Semaglutide for Weight Management in Subjects With Obesity
Brief Title: A Research Study to Investigate How Well NNC0165-1875 in Combination With Semaglutide Works in People With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9775-4708; U1111-1254-9046 (Other: WHO)
Record Dates: First submitted 2021-07-09; First posted 2021-07-21 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Part 1: is a 16-week study were one group of participants will receive two doses of NNC0165-1875 a week, in combination with one injection dose of semaglutide a week. The other group will receive a placebo.
  Part 2: is a 40-week study were one group of participants will receive one dose of NNC0165 a week, in combination with one injection dose of semaglutide a week. The other group will receive a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Semaglutide 2.4 mg and NNC0165-1875 2.0 mg (Experimental): Participants will receive two doses of NNC0165-1875 as an add on to semaglutide s.c. 2.4 mg
  Interventions: Drug: Semaglutide 2.4 mg and NNC0165-1875 2.0 mg
- Semaglutide 2.4 mg and placebo 2.0 mg(NNC0165-1875 2.0 mg) (Placebo Comparator): Participants will receive placebo as an add on to semaglutide 2.4 mg.
  Interventions: Drug: Semaglutide 2.4 mg and placebo 2.0 mg
- Semaglutide 2.4 mg and NNC0165-1875 1.0 mg (Experimental): Participants will receive two doses of NNC0165-1875 as an add on to semaglutide s.c. 2.4 mg
  Interventions: Drug: Semaglutide 2.4 mg and NNC0165-1875 1.0 mg
- Semaglutide 2.4 mg and placebo 1.0 mg(NNC0165-1875 1.0 mg) (Placebo Comparator): Participants will receive placebo as an add on to semaglutide 2.4 mg.
  Interventions: Drug: Semaglutide 2.4 mg and placebo 1.0 mg

INTERVENTIONS:
Drug: Semaglutide 2.4 mg and NNC0165-1875 2.0 mg — NNC0165-1875 will be co-escalated once-weekly subcutaneously with semaglutide every 2 weeks for the first 4 weeks, and every 4 weeks for the next 8 weeks until final target dose levels are reached.
  Arms: Semaglutide 2.4 mg and NNC0165-1875 2.0 mg
Drug: Semaglutide 2.4 mg and placebo 2.0 mg — NNC0165-1875 placebo will be co-escalated subcutaneously once-weekly with semaglutide every 2 weeks for the first 4 weeks, and every 4 weeks for the next 8 weeks until final target dose levels are reached.
  Arms: Semaglutide 2.4 mg and placebo 2.0 mg(NNC0165-1875 2.0 mg)
Drug: Semaglutide 2.4 mg and NNC0165-1875 1.0 mg — NNC0165-1875 will be co-escalated subcutaneously once-weekly with semaglutide every 2 weeks for the first 4 weeks, and every 4 weeks for the next 8 weeks until final target dose levels are reached.
  Arms: Semaglutide 2.4 mg and NNC0165-1875 1.0 mg
Drug: Semaglutide 2.4 mg and placebo 1.0 mg — NNC0165-1875 placebo will be co-escalated subcutaneously once-weekly with semaglutide every 2 weeks for the first 4 weeks, and every 4 weeks for the next 8 weeks until final target dose levels are reached.
  Arms: Semaglutide 2.4 mg and placebo 1.0 mg(NNC0165-1875 1.0 mg)

SUMMARY:
The study is looking at a new medicine to help people lose weight. In this study participants will either get semaglutide and NNC0165-1875 or semaglutide and a "dummy" medicine (placebo). Which treatment participants get is decided by chance. Participants will get 2 injections per week, on the same day. Participants will have to take the study medicine by use of a pre-filled pen. A pen is a medical tool with a needle used for injections under the skin. The study doctor or staff will show participants how. The study will last for about 26 weeks. Participants will have 17 visits at the clinic with the study doctor. At 4 of the clinic visits participants cannot eat and drink (water is allowed until 2 hours prior to the visit) for 8 hours before the visit.Women: Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period. Women who are able to become pregnant can participate if they agree to use contraception during the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* BMI 30.0-45.0 kg/m^2 (both inclusive) at the screening visit.

Exclusion Criteria:

* HbA1c greater than or equal to 48 mmol/mol (6.5%) as measured by a central laboratory at screening.

  * History of type 1 or type 2 diabetes mellitus.
  * Treatment with glucose-lowering agent(s) within 90 days before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (25):
- United States (25):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Profil Institute For Clinical Research Inc, Chula Vista, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Endo Res Solutions Inc, Roswell, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Altasciences Clinical Kansas, Inc., Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - AMC Community Endocrinology, Albany, New York
  - NYC Research, Inc., New York, New York
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Medical Uni of SC Charleston, Charleston, South Carolina
  - Coastal Carolina Res Ctr., North Charleston, South Carolina
  - Texas Diabetes & Endocrinology, P.A._Austin, Austin, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Texas Diabetes & Endocrinology, P.A._Austin, Round Rock, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Health Res of Hampton Roads, Newport News, Virginia
  - National Clin Res Inc., Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 14 sites in the United States.
Pre-assignment Details: The trial consisted of part 1 and 2. Part 1: 24 weeks (16-week treatment + 8 week follow up). In part 1 participants received NNC0165-1875 1.0 milligrams (mg) / matching placebo or NNC0165-1875 2.0 mg / matching placebo with semaglutide 2.4 mg. Part 2 further consisted of open-label run-in part (part 2a) of 32 weeks where participants received semaglutide and part 2b of 16 weeks where participants received NNC0165-1875 or NNC0165-1875 placebo with semaglutide s.c. 2.4 mg and 8-week follow up.
Groups:
- Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg: Participants received once-weekly subcutaneous (s.c) injection of NNC0165-1875 in a dose escalation manner (week 0-2: 0.05 mg, week 2-4: 0.1 mg, week 4-8: 0.25 mg, week 8-12: 0.5 mg, week 12 -16: 1.0 mg) along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 0-2: 0.25 mg, week 2-4: 0.5 mg, week 4-8: 1.0 mg, week 8-12: 1.7 mg, week 12 -16: 2.4 mg).
- Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 in a dose escalation manner (week 0-2: 0.1 mg, week 2-4: 0.25 mg, week 4-8: 0.5 mg, week 8-12: 1.0 mg, week 12 -16: 2.0 mg) along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 0-2: 0.25 mg, week 2-4: 0.5 mg, week 4-8: 1.0 mg, week 8-12: 1.7 mg, week 12 -16: 2.4 mg).
- Part 1: Placebo + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 matching placebo along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 0-2: 0.25 mg, week 2-4: 0.5 mg, week 4-8: 1.0 mg, week 8-12: 1.7 mg, week 12 -16: 2.4 mg).
- Part 2a (Run-in Period): Semaglutide 2.4 mg: Participants received once-weekly s.c injection of semaglutide in a dose escalation manner (week 0-2: 0.25 mg, week 2-4: 0.5 mg, week 4-6: 1.0 mg, week 6-8: 1.7 mg, week 8 -32: 2.4 mg). At week 32, participants who reached the target dose of semaglutide s.c. 2.4 mg and fulfilled the randomisation criteria entered Part 2b and randomised to receive either once-weekly NNC0165-1875 1.0 mg/ 2.0 mg or placebo along with once-weekly semaglutide 2.4 mg.
- Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 in a dose escalation manner (week 32-34: 0.05 mg, week 34-36: 0.1 mg, week 36-38: 0.25 mg, week 38-40: 0.5 mg, week 40 -48: 1.0 mg) along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 32-34: 0.25 mg, week 34-36: 0.5 mg, week 36-38: 1.0 mg, week 38-40: 1.7 mg, week 40-48: 2.4 mg).
- Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 in a dose escalation manner (week 32-34: 0.05 mg, week 34-36: 0.1 mg, week 36-38: 0.25 mg, week 38-40: 0.5 mg, week 40 -42: 1.0 mg, week 42-48: 2.0 mg,) along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 32-34: 0.25 mg, week 34-36: 0.5 mg, week 36-38: 1.0 mg, week 38-40: 1.7 mg, week 40-48: 2.4 mg).
- Part 2b: Placebo + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 matching placebo along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 32-34: 0.25 mg, week 34-36: 0.5 mg, week 36-38: 1.0 mg, week 38-40: 1.7 mg, week 40-48: 2.4 mg).
Period: Part 1 (24 Weeks)
Arm/Group | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 1: Placebo + Semaglutide 2.4 mg | Part 2a (Run-in Period): Semaglutide 2.4 mg | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Started | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2a: Run in Period (32 Weeks)
Arm/Group | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 1: Placebo + Semaglutide 2.4 mg | Part 2a (Run-in Period): Semaglutide 2.4 mg | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Started | 0 | 0 | 0 | 96 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 83 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 13 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2b (16 Weeks)
Arm/Group | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 1: Placebo + Semaglutide 2.4 mg | Part 2a (Run-in Period): Semaglutide 2.4 mg | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Started | 0 | 0 | 0 | 0 | 47 (Participants who achieved target dose of semaglutide 2.4 mg in Run in part randomized to Part 2b.) | 8 (Participants who achieved target dose of semaglutide 2.4 mg in Run in part randomized to Part 2b.) | 28 (Participants who achieved target dose of semaglutide 2.4 mg in Run in part randomized to Part 2b.)
Completed | 0 | 0 | 0 | 0 | 44 | 7 | 28
Not Completed | 0 | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants randomly assigned to trial treatment and who took at least one dose of trial product.
Groups:
- Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 in a dose escalation manner (week 0-2: 0.05 mg, week 2-4: 0.1 mg, week 4-8: 0.25 mg, week 8-12: 0.5 mg, week 12 -16: 1.0 mg) along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 0-2: 0.25 mg, week 2-4: 0.5 mg, week 4-8: 1.0 mg, week 8-12: 1.7 mg, week 12 -16: 2.4 mg).
- Part 2: All Participants randomised in Part 2.
- Total: Total of all reporting groups
Arm/Group | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 1: Placebo + Semaglutide 2.4 mg | Part 2 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 96 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44 (12) | 45 (14) | 43 (13) | 50 (13) | 48.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 78 | 91
  Male | 4 | 2 | 5 | 18 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 5 | 7
  Not Hispanic or Latino | 8 | 6 | 8 | 91 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 2
  Black or African American | 6 | 3 | 4 | 16 | 29
  White | 2 | 3 | 4 | 71 | 80
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an event that has onset after administration of trial product and no later than the follow-up visit or is present before trial product administration and increases in after the first dose of trial product and no later than the follow-up visit.
Time Frame: Part 1: From time of dosing (day 1) to follow-up (week 24)
Population: SAS included all participants randomly assigned to trial treatment and who took at least one dose of trial product This outcome measure is applicable for reported arms only.
Measure: Number; unit: Events
Arm/Group | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 1: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 8 | 8 | 8
Events | 56 | 71 | 37

2. Primary Outcome: Part 2b: Percentage Change in Body Weight
Description: Percentage change in body weight (%) from week 32 to week 48 is presented. For descriptive analysis and statistical analysis the endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2: Randomisation (week 32), end of treatment (week 48)
Population: Full analysis set (FAS) included all participants who were randomised. Overall number of participants analysed = Number of participants who contributed to the analysis. This outcome measure is applicable for reported arms only.
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Groups:
- Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg: Participants received once-weekly s.c injection of NNC0165-1875 in a dose escalation manner (week 32-34: 0.05 mg, week 34-36: 0.1 mg, week 36-38: 0.25 mg, week 38-40: 0.5 mg, week 40 -48: 1.0 mg) along with once-weekly s.c injection of semaglutide in a dose escalation manner (week 32-34: 0.25 mg, week 34-36: 0.5 mg, week 36-38: 1.0 mg, week 38-40: 1.7 mg, week 40-48: 2.4 mg).
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 44 | 26
Percentage change in body weight | -5.55 (3.97) | -3.06 (5.46)
Statistical Analysis 1: Comparison: Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg vs Part 2b: Placebo + Semaglutide 2.4 mg; Week 48 responses were analysed using an analysis of covariance model with randomised treatment as factors and baseline body weight (kg) as covariate; Test type: Superiority; p = 0.0437, ANCOVA; Treatment difference (%-point) = -2.15, 95% CI 2-sided [-4.24 to -0.06]

3. Secondary Outcome: Part 2b: Change in Body Weight (kg)
Description: Change in body weight (kg) from week 32 to week 48 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: FAS included all participants who were randomised. Overall number of participants analysed = Number of participants who contributed to the analysis. This outcome measure is applicable for reported arms only.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 44 | 26
kilograms (kg) | -4.54 (3.22) | -2.23 (5.16)

4. Secondary Outcome: Part 2b: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change in HbA1c from week 32 to week 48 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Percentage point is calculated by subtraction of baseline HbA1c from HbA1c at end of treatment.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 44 | 26
Percentage point of HbA1c | -0.17 (0.17) | -0.17 (0.14)

5. Secondary Outcome: Part 2b: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG (measured in millimoles per liter [mmol/l]) from week 32 to week 48 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: FAS included all partcipants who were randomised. Overall number of participants analysed = Number of participants who contributed to the analysis. This outcome measure is applicable for reported arms only.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 25
mmol/l | 0.08 (0.36) | -0.02 (0.42)

6. Secondary Outcome: Part 2b: Change in Fasting Insulin
Description: Change in fasting insulin (measured in picomoles per liter [pmol/l]) from week 32 to week 48 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 24
pmol/l | -14.10 (39.31) | -8.10 (47.22)

7. Secondary Outcome: Part 2b: Change in Waist Circumference
Description: Change in waist circumference (measured in centimeter [cm]) from week 32 to week 48 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 44 | 27
cm | -4.80 (6.92) | -2.69 (5.73)

8. Secondary Outcome: Part 2b: Relative Change in Total Cholesterol (Ratio to Baseline)
Description: Relative change in total cholesterol (measured in mmol/L) from week 32 to week 48 is presented as ratio to baseline. here baseline = Randomisation (week 32). The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of total cholesterol
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 23
Ratio of total cholesterol | 1.00 (0.11) | 1.07 (0.17)

9. Secondary Outcome: Part 2b: Relative Change in High Density Lipoprotein (HDL) Cholesterol (Ratio to Baseline)
Description: Relative change in HDL cholesterol (measured in mmol/L) from week 32 to week 48 is presented as ratio to baseline. here baseline = Randomisation (week 32). The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of HDL cholesterol
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 23
Ratio of HDL cholesterol | 1.02 (0.12) | 1.08 (0.12)

10. Secondary Outcome: Part 2b: Relative Change in Low Density Lipoprotein (LDL) Cholesterol (Ratio to Baseline)
Description: Relative change in LDL cholesterol (measured in mmol/L) from week 32 to week 48 is presented as ratio to baseline. here baseline = Randomisation (week 32). The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of LDL cholesterol
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 23
Ratio of LDL cholesterol | 1.01 (0.17) | 1.08 (0.27)

11. Secondary Outcome: Part 2b: Relative Change in Very Low Density Lipoprotein (VLDL) Cholesterol (Ratio to Baseline)
Description: Relative change in VLDL cholesterol (measured in mmol/L) from week 32 to week 48 is presented as ratio to baseline. here baseline = Randomisation (week 32). The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of VLDL cholesterol
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 23
Ratio of VLDL cholesterol | 0.96 (0.25) | 1.04 (0.27)

12. Secondary Outcome: Part 2b: Relative Change in Triglycerides (TG) (Ratio to Baseline)
Description: Relative change in triglycerides (measured in mmol/l) from week 32 to week 48 is presented as ratio to baseline. here baseline = Randomisation (week 32). The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of triglycerides
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 23
Ratio of triglycerides | 0.96 (0.26) | 1.03 (0.26)

13. Secondary Outcome: Part 2b: Relative Change in Free Fatty Acids (Ratio to Baseline)
Description: Relative change in free fatty acids (measured in mmol/L) from week 32 to week 48 is presented as ratio to baseline. here baseline = Randomisation (week 32). The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Part 2b: Randomisation (week 32), end of treatment (week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of free fatty acids
Arm/Group | Part 2b: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 43 | 25
Ratio of free fatty acids | 0.87 (0.39) | 1.07 (0.48)

14. Secondary Outcome: Part 2b: Number of Treatment -Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical trial participant that is temporally associated with the use of an IMP, whether or not considered related to the IMP. All AEs reported here are TEAEs. A TEAE is defined as an event that has onset after administration of trial product and no later than the follow-up visits or is present before trial product administration and increases in after the first dose of trial product and no later than the follow-up visit. The TEAEs occurred from week 32 to week 56 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: From randomisation (week 32) to end of the trial (week 56)
Population: SAS included all participants randomly assigned to trial treatment and who took at least one dose of trial product. This outcome measure is applicable for reported arms only.
Measure: Number; unit: Events
Arm/Group | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 47 | 8 | 28
Events | 220 | 45 | 56

15. Secondary Outcome: Part 2b: Number of Treatment-emergent Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. The SAEs occurred from week 32 to week 56 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: From randomisation (week 32) to end of the trial (week 56)
Population: as for outcome 14
Measure: Number; unit: Events
Arm/Group | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
Number analyzed (Participants) | 47 | 8 | 28
Events | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From week 0 to week 80 (Part 1: week 0 to follow-up (week 24); Part 2: From baseline at (week 0) to end of trial (week 56) Results are based on the SAS included all participants randomly assigned to trial treatment and who took at least one dose of trial product.
Description: All AEs reported here are TEAEs. A TEAE is defined as an event that either has onset after administration of trial product and no later than the follow-up visit. SAS included all participants randomly assigned to trial treatment and who took at least one dose of trial product.
Arm/Group | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 1: Placebo + Semaglutide 2.4 mg | Part 2a (Run-in Period): Semaglutide 2.4 mg | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg | Part 2b: Placebo + Semaglutide 2.4 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/96 | 0/47 | 0/8 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/8 | 2/96 | 2/47 | 0/8 | 0/28
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 69/96 | 36/47 | 7/8 | 16/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg (N=8) | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg (N=8) | Part 1: Placebo + Semaglutide 2.4 mg (N=8) | Part 2a (Run-in Period): Semaglutide 2.4 mg (N=96) | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg (N=47) | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg (N=8) | Part 2b: Placebo + Semaglutide 2.4 mg (N=28)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: NNC0165-1875 1.0 mg + Semaglutide 2.4 mg (N=8) | Part 1: NNC0165-1875 2.0 mg + Semaglutide 2.4 mg (N=8) | Part 1: Placebo + Semaglutide 2.4 mg (N=8) | Part 2a (Run-in Period): Semaglutide 2.4 mg (N=96) | Part 2b : NNC0165-1875 1.0 mg + Semaglutide 2.4 mg (N=47) | Part 2b : NNC0165-1875 2.0 mg + Semaglutide 2.4 mg (N=8) | Part 2b: Placebo + Semaglutide 2.4 mg (N=28)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (7) | 6 (6) | 5 (5) | 2 (2) | 2 (2) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early Satiety (General disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Reaction (General disorders) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular Filtration Rate Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Taste Disorder (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood Swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (3) | 0 (0) | 1 (1) | 4 (9) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 18 (19) | 12 (12) | 4 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 16 (20) | 5 (8) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 3 (3) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (3) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (9) | 1 (1) | 39 (50) | 21 (39) | 5 (8) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (6) | 6 (8) | 0 (0) | 16 (21) | 15 (34) | 3 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Transient lingual papillitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 8 (9) | 4 (10) | 0 (0) | 1 (3)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (2) | 5 (5) | 1 (1) | 8 (8) | 1 (1) | 1 (2) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 17 (17) | 4 (4) | 0 (0) | 3 (3)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04969939/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04969939/SAP_001.pdf